CLINICAL TRIAL: NCT00847535
Title: Muscle Cell Mediated Therapy for Stress Urinary Incontinence: An Investigation of the Safety of 4 Different Doses of Autologous Muscle Derived Cells.
Brief Title: An Investigation of the Safety of 4 Different Doses of Autologous Muscle Derived Cells as Therapy for Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cook MyoSite (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-006; IND1
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2014-01-01 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Stress Urinary Incontinence; Cell Therapy
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (2):
- 1 (Other): Transurethral dose escalation
  Interventions: Biological: autologous muscle cell injection
- 2 (Other): Periurethral dose escalation
  Interventions: Biological: autologous muscle cell injection

INTERVENTIONS:
Biological: autologous muscle cell injection — Injection of autologous muscle cells

SUMMARY:
This is a clinical investigation approved by US FDA and Canadian Health Authority to study the safety and potential effectiveness of the autologous muscle cells for the treatment of stress urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Patient has SUI with normal detrusor activity confirmed with urodynamics
* Patient has bladder capacity >200 mL
* Patient's incontinence has not shown any improvement for at least -6 months
* Patient has failed prior treatments (e.g., behavior modification, bladder exercises, biofeedback, electrical stimulation, bulking injections, urethral suspensions and/or drug therapy)

Exclusion Criteria:

* Patient has known vesicoureteral reflux, vaginal prolapse beyond the introitus, or other significant pelvic floor abnormalities with high pressure instability
* Patient has a neuromuscular disorder (e.g., muscular dystrophy, multiple sclerosis)
* Patient has uncontrolled diabetes
* Patient is pregnant, lactating, or plans to become pregnant during the course of the study
* Patient is morbidly obese (defined as 100 pounds over their ideal body weight, or BMI ≥40) and would not be expected to benefit from treatment
* Patient has current or acute conditions involving cystitis or urethritis
* Patient is scheduled to receive radiation treatment to the vicinity
* Patients with a history of radiation treatment to the urethra or adjacent structures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-10-09 (Actual); Primary Completion 2011-11-02 (Actual); Study Completion 2011-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (3):
- United States (2):
  - Wm Beaumont Hospital, Royal Oak, Michigan
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada

REFERENCES:
- See also: Autologous muscle derived cells for treatment of stress urinary incontinence in women — http://www.ncbi.nlm.nih.gov/pubmed/24582537

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 66 participants were biopsied, 64 participants received injections.
Groups:
- Part I: Transurethral Injection; Part I: Periurethral Injection; Part II: Transurethral Injection: Autologous Muscle-Derived Cells (AMDC) are intended for use in the treatment of stress urinary incontinence (SUI) in women. Following skeletal muscle biopsy of the thigh to obtain starting material for production of AMDC, patients underwent intrasphincteric injection of AMDC.
Period: Overall Study
Arm/Group | Part I: Transurethral Injection | Part I: Periurethral Injection | Part II: Transurethral Injection
Started | 24 | 24 | 16
10 Million AMDC | 8 | 8 | 0
50 Million AMDC | 8 | 8 | 0
100 Million AMDC | 8 | 8 | 8
200 Million AMDC | 0 | 0 | 8
Completed | 22 | 22 | 15
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Treated With AMDC: Autologous Muscle-Derived Cells (AMDC) are intended for use in the treatment of stress urinary incontinence (SUI) in women.
Arm/Group | Patients Treated With AMDC
Number analyzed (Participants) | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Biopsy Procedure-related Adverse Events
Description: Biopsy was required to generate AMDC products. Biopsy procedure-related events were defined as systemic responses to the biopsy procedure or injury at the biopsy site. Since biopsy occurred prior to AMDC treatment, results are presented independent of AMDC dose received.
  All biopsy procedure-related events either self-resolved or were easily treated.
Time Frame: at biopsy or between biopsy and treatment
Population: During the study, 66 patients underwent a total of 78 biopsies.
Measure: Number; unit: participants
Groups:
- Patients With Biopsy: Autologous Muscle-Derived Cells (AMDC) are intended for use in the treatment of stress urinary incontinence (SUI) in women.
Arm/Group | Patients With Biopsy
Number analyzed (Participants) | 66
participants | 3

2. Primary Outcome: Biopsy Procedure-related Adverse Events
Description: as for outcome 1
Time Frame: at biopsy or between biopsy and treatment
Measure: Number; unit: Number of events
Arm/Group | Patients With Biopsy
Number analyzed (Participants) | 66
Number of events
  Wound hematoma | 2
  Post procedural hemorrhage | 1
  Joint swelling | 1
  Feeling hot | 1
  Procedural dizziness | 1
  Hyperhidrosis | 1

3. Primary Outcome: Number of Participants That Experienced Injection Procedure-related Adverse Events
Description: AMDC treatment was administered via intrasphincteric injection. Injection procedure-related events were defined as systemic responses to the injection procedure or genitourinary events occurring within 30 days of the injection procedure that could be attributed to cystoscopy or catheterization. Since these events could be attributed to the injection procedure, results are considered independent of AMDC dose received.
  All injection procedure-related events self-resolved or were easily treated.
Time Frame: 30 days
Population: Sixty-four patients underwent intrasphincteric injection of AMDC.
Measure: Number; unit: participants
Arm/Group | Patients Treated With AMDC
Number analyzed (Participants) | 64
participants | 8

4. Primary Outcome: Injection Procedure-related Adverse Events
Description: as for outcome 3
Time Frame: 30 days
Measure: Number; unit: Number of events
Arm/Group | Patients Treated With AMDC
Number analyzed (Participants) | 64
Number of events
  Dysuria | 3
  Vulvovaginal pruritis | 3
  Pelvic/abdominal pain | 2
  Hematuria | 2
  Vulvovaginal burning sensation | 1
  Sensation of foreign body | 1
  Pollakiuria | 1
  Micturition urgency | 1

5. Primary Outcome: Number of Participants That Experienced AMDC Product-related Adverse Events
Description: If an immune response after injection or any urinary retention occurred and seemed suspicious, the physicians were consulted to determine whether the effect was likely related to the AMDC product.
  No adverse events reported during the study were adjudicated as AMDC product-related.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Patients Treated With AMDC
Number analyzed (Participants) | 64
participants | 0

ADVERSE EVENTS:
Time Frame: Biopsy to treatment, 12 months Post-treatment
Description: During the study, 66 patients underwent a total of 78 biopsies, and 64 patients underwent intrasphincteric injection of AMDC.
Groups:
- Patients: Autologous Muscle-Derived Cells (AMDC) are intended for use in the treatment of stress urinary incontinence (SUI) in women
Arm/Group | Patients
Serious Adverse Events (participants affected / at risk) | 8/66
Other Adverse Events (participants affected / at risk) | 18/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Patients (N=66)
Biopsy to treatment: Drug hypersensitiviy (Immune system disorders) | 1 (1)
Biopsy to treatment: Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Post-treatment: Angina unstable (Cardiac disorders) | 1/64 (1)
Post-treatment: Cardiac failure congestive (Cardiac disorders) | 1/64 (1)
Post-treatment: Enterocolitis infectious (Gastrointestinal disorders) | 1/64 (1)
Post-treatment: Intervertebral disc operation (Surgical and medical procedures) | 1/64 (1)
Post-treatment: Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1/64 (1)
Post-treatment: Myocardial infarction (Cardiac disorders) | 1/64 (1)
Post-treatment: Small intestinal obstruction (Gastrointestinal disorders) | 1/64 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Patients (N=66)
Biopsy to treatment: Urinary tract infection (Renal and urinary disorders) | 4 (4)
Post-treatment: Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4/64 (4)
Post-treatment: Dysuria (Renal and urinary disorders) | 5/64 (5)
Post-treatment: Pollakiuria (Renal and urinary disorders) | 4/64 (4)
Post-treatment: Urinary tract infection (Renal and urinary disorders) | 5/64 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days